CLINICAL TRIAL: NCT02508467
Title: A Phase 1 Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of BLU-554 in Patients With Hepatocellular Carcinoma
Brief Title: A Phase 1 Study of Fisogatinib (BLU-554) in Patients With Hepatocellular Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Blueprint Medicines Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BLU-554-1101; 2015-001662-26 (EudraCT Number)
Record Dates: First submitted 2015-07-09; First posted 2015-07-27 (Estimated); Last update posted 2024-04-12 (Actual); Status verified 2024-03

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Liver cancer; FGF19 gene amplification; FGF19 overexpression; FGF19 upregulation; Cyclin D1 (CCND1) gene amplification; Cyclin D1 (CCND1) copy number gain; BLU-554; FGFR4; Hepatocellular carcinoma; Liver Disease; Liver Neoplasms
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Liver Diseases | interventions — fisogatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fisogatinib (BLU-554) (Experimental): Fisogatinib (BLU-554) capsules for oral administration.
  Interventions: Drug: Fisogatinib (BLU-554)

INTERVENTIONS:
Drug: Fisogatinib (BLU-554)
  Other Names: BLU-554

SUMMARY:
This is a Phase 1, open-label, first-in-human (FIH) study designed to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary antineoplastic activity of fisogatinib (formerly known as BLU- 554) administered orally in patients with FGF19 IHC+ hepatocellular carcinoma (HCC). The study consists of 3 parts, a dose-escalation part (Part 1), an expansion part (Part 2) exploring a once daily (qd) dosing schedule at the recommended Phase 2 dose (RP2D), and a Part 3 expansion of the qd dosing schedule at the RP2D in TKI naive patients.

ELIGIBILITY:
Key Inclusion Criteria:

* Confirmed diagnosis of HCC by histological examination or by non-invasive criteria according to European Association for the Study of the Liver (EASL) or American Association for the Study of Liver Disease (AASLD) guidelines (Part 1, 2 and 3).
* For Part 1 and 2, the patient has unresectable disease and has been previously treated with sorafenib, has declined treatment with sorafenib, or does not have access to sorafenib.
* For Part 3, the patient has not received prior treatment with a TKI.
* Child-Pugh class A with no clinically apparent ascites
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* For Part 1, willing to provide archived tumor tissue (if available) and willing to undergo pre- and on-treatment tumor biopsy (if considered safe and medically feasible by the treating investigator)
* For Part 2 and 3, all patients must have an FGF19 IHC result available. Only FGF19 IHC+ HCC patients will be eligible for Part 3.

Key Exclusion Criteria:

* Central nervous system metastases
* Platelet count <75,000/mL
* Absolute neutrophil count <1000/mL
* Hemoglobin <8 g/dL
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >5x the upper limit of normal (ULN)
* Total bilirubin >2.5 mg/dL
* International normalized ratio (INR) >2.3 or prothrombin time (PT) >6 seconds above control
* Estimated (Cockroft-Gault formula) or measured creatinine clearance <40 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2015-07-31 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) on qd and bid schedules | During cycle 1 (28 days) of treatment and will be determined by approximately 24 months after start of the study or earlier
Recommended Phase 2 dose of fisogatinib (BLU-554) on qd and bid schedules | At the end of every cycle (28 days) of treatment and will be determined by approximately 24 months after start of the study or earlier
Number of patients with adverse events, serious adverse events and changes in physical findings, vital signs, clinical laboratory results and ECG findings | Every cycle (28 days) for approximately 24 months or earlier if patient terminates from the study

SECONDARY OUTCOMES:
Maximum plasma concentration of fisogatinib (BLU-554) on qd and bid schedules | Every cycle (28 days) up to cycle 4 and at end of treatment (approximately 24 months or earlier if patient terminates from the study)
  Blood samples may be taken at pre-dose, and 0.5, 1, 2, 4, 6, 8 and 24 hrs post dose on Cycle 1 Day 1 and Cycle 1 Day 15, Pre-dose of Cycle 2 to 4, Day 1 and end of treatment (EOT)
Time to maximum plasma concentration of fisogatinib (BLU-554) on qd and bid schedules | Every cycle (28 days) up to cycle 4 and at end of treatment (approximately 24 months or earlier if patient terminates from the study)
  Blood samples may be taken at pre-dose, and 0.5, 1, 2, 4, 6, 8 and 24 hrs post dose on Cycle 1 Day 1 and Cycle 1 Day 15, Pre-dose of Cycle 2 to 4, Day 1 and EOT
Fibroblast growth factor 19 (FGF19) status in tumor tissue | Cycle 2 (Day 56)
Levels of FGF19 in blood and tumor samples | Cycle 1 (Day 28)
Preliminary evidence of fisogatinib (BLU-554) antineoplastic activity | Screening, Day 1 of every odd numbered cycle starting with Cycle 3, End of treatment (at approximately 24 months or earlier if patient terminates from the study) and every three months post EOT

CONTACTS AND LOCATIONS:
Locations (41):
- United States (7):
  - Inland Empire Liver Foundation, Rialto, California
  - University of Miami - Sylvester Comprehensive Cancer Center, Miami, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Ochsner Cancer Institute, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai Medical Center, New York, New York
  - Huntsman Cancer Institute, Salt Lake City, Utah
- China (14):
  - Zhejiang Cancer Hospital, Hangzhou, Gongshu District
  - Nanfang Hospital, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Radioactive Interventional Department, Changsha, Hunan
  - The Chinese People's Liberation Army 81 Hospital, Nanjing, Jiangsu
  - Nantong Tumor Hospital, Nantong, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - Jilin University the First Affiliated Hospital, Changchun, Jilin
  - Fudan University Zhongshan Hospital, Xuhui, Shanghai City
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Hepatobiliary Oncology Department, Tianjin, West Lake District
  - Fudan University Shanghai Cancer Center, Shanghai, Xuhui District
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
- France (2):
  - Hospital Beaujon, Clichy
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Johannes Gutenberg University Mainz - University Medical Center, Mainz, Rhineland-Palatine
  - University of Frankfurt, Frankfurt
- Hong Kong (2):
  - Prince of Wales Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- IRCCS Foundation - National Institute of Tumors, Milan, Italy
- National Cancer Centre, Singapore, Singapore
- South Korea (4):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Vall d'Hebron Institute of Oncology, Barcelona, Spain
- Inselspital Bern, Bern, Switzerland
- Taiwan (2):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- United Kingdom (4):
  - University of Liverpool - Clatterbridge Cancer Centre, Bebington
  - Royal Free Hospital, London
  - Guy's Hospital, London
  - University College London, London